CLINICAL TRIAL: NCT00003269
Title: A Phase II, Open-Label, Trial Evaluating the Efficacy of Amifostine in Patients With Cancers Receiving Outpatient Dose-intensive Cyclophosphamide, Etoposide, and Cisplatin (DICEP) Chemotherapy
Brief Title: Amifostine Followed by High Dose Chemotherapy in Treating Patients With Hematologic Cancer or Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: James R. Mason, M.D., Scripps Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000066165; SCRF-98014 (Other: Scripps Health); ALZA-97-49-ii (Other: Alza Corporation); NCI-V98-1396 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer; Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Lymphoma; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIB breast cancer; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; Waldenstrom macroglobulinemia; limited stage small cell lung cancer; extensive stage small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; drug/agent toxicity by tissue/organ; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Lymphoma; Ovarian Neoplasms; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Lymphoma, T-Cell, Cutaneous; Carcinoma, Ovarian Epithelial; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — sargramostim; Amifostine; Cisplatin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: sargramostim
Drug: amifostine trihydrate
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Randomized phase II trial to study the effectiveness of amifostine followed by high-dose chemotherapy in treating patients with hematologic cancer or solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of amifostine in enhancing hematopoietic recovery following cyclophosphamide, etoposide, and cisplatin therapy in patients with hematologic malignancies and adult solid tumors.

OUTLINE: This is an open label study. Patients receive intravenous amifostine over 15 minutes daily 30 minutes prior to high dose chemotherapy on days 0-2. Cyclophosphamide is administered over 3 hours on days 0 and 1, intravenous etoposide over 4 hours on days 0, 1, and 2, and cisplatin over 4 hours on days 0, 1, and 2. All patients receive sargramostim (GM-CSF) beginning on day 4. Patients receive a maximum of 2 courses of treatment (with 35-42 days between chemotherapy courses). Patients are followed for 1-5 months after treatment.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hematologic malignancies and adult solid tumors, including: Non-Hodgkin's lymphoma Lung cancer Hodgkin's disease Ovarian cancer Breast cancer No refractory disease (less than partial response to induction chemotherapy) No CNS metastases No unilateral bone marrow biopsy within 6 months of study showing at least 20% involvement by fibrosis tumors Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 70 Menopausal status: Not specified Performance Status: ECOG 0-2 Life expectancy: At least 16 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT or SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2 mg/dL Other: HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No underlying medical or psychiatric conditions No concurrent active infection No prior malignancies except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior myeloid growth factor Chemotherapy: At least 4 weeks since prior chemotherapy No more than 1 prior chemotherapy regimen (excluding adjuvant chemotherapy) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since pelvic, para-aortic, inverted Y, cranial, spinal, or mediastinal radiation Surgery: At least 2 weeks since major surgery Other: No antihypertensive medication within 24 hours of amifostine administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1998-02; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
duration of neutropenia | 30 days
  number of days absolute neutrophil count less than 500 during the nadir period after administration of high dose chemotherapy

SECONDARY OUTCOMES:
incidence of nephrotoxicity | 30 days
  decrease in creatinine clearance from baseline after high dose chemotherapy
incidence of ototoxicity | 30 days
  change in audiogram from baseline after high dose chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: James R. Mason, MD, Study Chair — Ida M. and Cecil H. Green Cancer Center at Scripps Clinic
Locations (1):
- Scripps Clinic, La Jolla, California, United States